CLINICAL TRIAL: NCT05173727
Title: Prevalence and Serotype of Streptococcus Pneumoniae in Hospitalized Adult With Community-Acquired Pneumonia: Isolated From Blood, Nasopharyngeal Swab, Urine, and/or Sputum
Brief Title: Prevalence and Serotype of Streptococcus Pneumoniae Hospitalized Adult With Community-Acquired Pneumonia
Acronym: HACAP
Status: Completed | Type: Observational
Sponsor: Dr Cipto Mangunkusumo General Hospital (Other)
Collaborators: Eijkman Institute for Molecular Biology (Other)
Responsible Party: Principal Investigator, Gurmeet Singh, MD, Head Division Respirology and Critical Illness, Internal Medicine Department, Principal Investigator, Respirology and Critical Illness Consultant, Dr Cipto Mangunkusumo General Hospital
Other Study IDs: 61356
Record Dates: First submitted 2021-12-10; First posted 2021-12-30 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-11

CONDITIONS: Pneumonia, Bacterial
MeSH Terms: conditions — Pneumonia, Bacterial

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Streptococcus Pneumoniae is one of the etiology in severe CAP and accounts for about 60-75% of cases and is likely to be the leading cause of unknown etiologic pneumonia. In Indonesia, studies regarding the prevalence of Streptococcus pneumoniae as the cause of CAP are still very rare. Therefore, there is still a need for further investigation in S. pneumoniae prevalence among hospitalized CAP by utilizing different detection methods in Indonesia. Antibiotics as a therapy of CAP also showed high levels of resistance, meanwhile, early detection of causative pathogen is potentially reducing the incidence of antibiotic resistance and usage of broad-spectrum antibiotics.

DETAILED DESCRIPTION:
Pneumonia is inflammation of the lungs by bacteria with symptoms of high fever accompanied by productive cough, rapid breathing (frequency of breath >50 times/minutes), tightness, and other symptoms (headache, restlessness, and reduced appetite). Pneumonia is a health problem in the world due to high morbidity and mortality. Streptococcus pneumoniae is one of the etiology in severe community-acquired pneumonia (CAP) and accounts for about 60-75% of cases and is likely to be the leading cause of unknown etiologic pneumonia. In Indonesia, studies regarding the prevalence of Streptococcus pneumoniae as the cause of CAP are still very rare. Previous study (Amanda,2020) found that Streptococcus pneumoniae prevalence isolated from CSF and blood in adult CAP patients is very low (around 14% from 100 patients). Therefore, there is still a need for further investigation in S. pneumoniae prevalence among hospitalized CAP by utilizing different detection methods in Indonesia.

Diagnosis relies upon microbiological confirmation of Streptococcus pneumoniae in patients with clinical and radiological features of pneumonia. Blood culture remains the gold standard for confirmation of Streptococcus pneumoniae and only occurs in 15-30% of cases. Furthermore, treatment with antibiotics before specimen sampling reduces the sensitivity in the majority of the cases. Urine antigen detection is a non-invasive test to detect C polysaccharide antigen in urine has good sensitivity and very specific in the adult patient with Streptococcus pneumoniae infection. A meta-analysis and systematic review in 2013 mentioned the sensitivity value of urine-based pneumococcal antigen reached 67.6% (CI 95%) and specificity 98.1% (CI 95%). In addition, a study by Molinos et al. (2015) found out that 21% of all caused CAP patients are positive with S. pneumoniae detected by urine antigen test.

Antibiotics as a therapy of CAP showed high levels of resistance. Yu et al (2011) reported Streptococcus pneumoniae as the main cause of community-acquired pneumonia has been resistance to antibiotics of penicillin (in vitro), macrolides, and quinolones. Early detection of the causative pathogen can reduce the incidence of antibiotic resistance and the usage of broad-spectrum antibiotics.

To investigators' knowledge, this study will be the first to assess and evaluate multiple methods for the detection of S. pneumoniae by collecting and testing respiratory and non-respiratory samples from the hospitalized adult with CAP in Indonesia.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized adult ≥ 18 years old
* Moderate to severe CAP (CURB-65 score > 2 dan ATS/IDSA 2019)

Exclusion Criteria:

* Have been taking antibiotic more than 24 hours before enrollment.
* Diagnose with non-infectious ARDS disease (such as aspiration pneumonia or cardiogenic pulmonary edema).
* Diagnose with tuberculosis based on clinical or radiological findings.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population target is the severe pneumonia patient in ED/ICU/HCU Cipto Mangunkusumo Hospital. The reachable population is moderate and severe CAP in ED/ICU/HCU, Cipto Mangunkusumo Hospital., Jakarta. The research subjects are the reachable population who meet the inclusion and exclusion criteria by consecutive sampling recruitment method
Sampling Method: Non-Probability Sample
Enrollment: 355 (Actual)
Dates: Start 2022-05-15 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Determine the distribution of Streptococcus pneumoniae serotype and its prevalence | Through study completion, an average of 2 year.
  Determine the distribution of Streptococcus pneumoniae serotype and its prevalence isolated from hospitalized adult patients with CAP in Cipto Mangunkusumo Hospital, Jakarta, Indonesia utilizing different methods.

SECONDARY OUTCOMES:
To investigate the antibiotics susceptibility of Streptococcus pneumoniae | Through study completion, an average of 2 year
  To investigate the antibiotics susceptibility of Streptococcus pneumoniae in hospitalized adult patients with CAP

CONTACTS AND LOCATIONS:
Overall Officials: Gurmeet Singh, MD, PhD, Principal Investigator — Indonesian Society of Respirology
Locations (1):
- Cipto Mangunkusumo Hospital - Universitas Indonesia, Jakarta Pusat, Jakarta Special Capital Region, Indonesia

IPD SHARING:
Plan to Share IPD: No